CLINICAL TRIAL: NCT05237908
Title: Prospective, Randomized, Single-Blind Study for the Evaluation of the Clinical Outcome and the Fusion Rate of 3D Printed Interbody Fusion Cages and Titanium Coated PEEK Cages in Transforaminal Lumbar Interbody Fusion
Brief Title: Clinical Outcome and Fusion Rate of 3D Printed Interbody Fusion Cages and Titanium Coated PEEK Cages
Acronym: PRINTLIF
Status: Active, not recruiting | Type: Observational
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-2114
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Disk Herniated Lumbar; Disc Disease Degenerative; Spondylolisthesis
Keywords: Transforaminal lumbar interbody fusion
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spondylolisthesis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TSPACE 3D: the 3D printed cage (TSPACE 3D) is defined as investigational product
  Interventions: Device: Transforaminal Lumbar Interbody Fusion
- TSPACE XP: the titanium coated PEEK cage (TSPACE XP) is defined as reference product.
  Interventions: Device: Transforaminal Lumbar Interbody Fusion

INTERVENTIONS:
Device: Transforaminal Lumbar Interbody Fusion — Interbody Fusion means the operative immobilization or ankylosis of two or more vertebrae by fusion of the vertebral bodies with a short bone graft or often with diskectomy or laminectomy. (From Blauvelt and Nelson, A Manual of Orthopaedic Terminology, 5th ed, p236; Dorland, 28th ed

SUMMARY:
Prospective, Randomized, Single-Blind Study for the Evaluation of the Clinical Outcome and the Fusion Rate of 3D Printed Interbody Fusion Cages and Titanium Coated PEEK Cages in Transforaminal Lumbar Interbody Fusion

DETAILED DESCRIPTION:
This clinical study is a regulatory Post Market Clinical Follow-Up (PMCF) measure and is aiming to collect clinical data on the performance and safety of the TSPACE® 3D implants. It is designed as a prospective, randomized, single-blind, non-interventional study in order to gain clinical data within the routine clinical application of the investigational device.

The study shall answer the question if there are detectable differences between the established titanium coated Polyether Ether Ketone (PEEK) cages of the manufacturer and the new 3D printed cages. Differences shall be observed in terms of clinical outcome, quality of life, patient satisfaction, radiological outcome and occurrence of Adverse Events / Serious Adverse Events.

ELIGIBILITY:
Inclusion Criteria:

* Indication for one, two or three-segment lumbar interbody fusion according to Instructions for use
* Written informed consent for the documentation of clinical and radiological results
* Willingness and mental ability to participate at the follow-up examinations

Exclusion Criteria:

* Patient is not willing or able to participate at the follow-up examination
* Patient age < 18 years and >80 years
* Patient is pregnant
* Previous instrumented lumbar spine surgery

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited consecutively. No selection besides the inclusion and exclusion criteria will take place.
Sampling Method: Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2022-02-18 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Clinical outcome measured with the Oswestry Disability Index | 1 year postoperatively
  The Oswestry Disability Index is designed to measure back-specific disability. The questionnaire is self-administered and has 10 items concerning pain and activities of daily living including personal care, lifting, walking, sitting, standing, sleeping, sex life, social life and travelling. It is a self-administered questionnaire Each section is scored on a 0-5 scale, 5 is for maximum disability. The index is calculated by dividing the total score by the total possible score, which is multiplied by 100 and expressed as a percentage. The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.

SECONDARY OUTCOMES:
Clinical improvement: pain | preoperatively, at 3 months, 1 year, 2 years and 5 years postoperatively
  Pain will be assessed by the patient using the Visual Analogue Scale (VAS) which state "0" at one end representing "no pain" and "100" at the opposite end representing "maximal/worst pain"
Development Quality of life (EQ-5D-5L) | preoperatively, at 3 months, 1 year, 2 years and 5 years postoperatively
  EQ-5D-5L is a standardized 5-dimension 5-level measure of the health status and is developed by the EuroQol Group in order to have a simple and generic measure for clinical and economic assessment. In order to analyze the quality of life of the patients, the EQ-5D-5L is used. The score is self-completed by the patient and will therefore be used in German.
Radiological outcome: Fusion | 1 year postoperatively
  Bone fusion: After interbody fusion surgery fusion of the treated segment is aspired. Thus, the implant design shall allow on-/ingrowth to/into the material. The fusion status can be determined from radiographs (static or dynamic). Bony fusion can be characterized quantitatively by the fusion rate.
Radiological outcome: Implant subsidence | 1 year postoperatively
  Implant penetration into the vertebral body occurs frequently after spinal reconstruction. Interbody fusion cages may subside into the vertebral body and lead to kyphotic deformity
Radiological outcome: Implant migration | 1 year postoperatively
  Interbody fusion cages might migrate forward into the retroperitoneum or backwards into the vertebral canal and can, thus, cause serious clinical consequences (e.g. compression of nerve roots or dura mater).
Rate of (Serious) adverse events | throughout the studies duration up to five years postoperatively
  Occurrence of complications potentially associated with the implanted devices can never be fully excluded during spinal surgery. In order to monitor potential complication and to identify so far unknown complications adverse events (AE) and serious adverse events (SAE) deemed related to the investigational device are recorded.
Development of Clinical outcome measured with the Oswestry Disability Index | preoperatively, at 3 months, 1 year, 2 years and 5 years postoperatively.
  The Oswestry Disability Index is designed to measure back-specific disability. The questionnaire is self-administered and has 10 items concerning pain and activities of daily living including personal care, lifting, walking, sitting, standing, sleeping, sex life, social life and travelling. It is a self-administered questionnaire Each section is scored on a 0-5 scale, 5 is for maximum disability. The index is calculated by dividing the total score by the total possible score, which is multiplied by 100 and expressed as a percentage. The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.

OTHER OUTCOMES:
Duration of surgery | Intraoperative
  Duration of the intervention from first cut to suturing
Blood loss | intraoperative
  Amount of Blood loss due to the intervention
Length of hospital stay | up to patient's discharge from hospital (approximately 5 days postoperatively)
  Number of days the patient has to stay in hospital after the intervention
Development of Patient satisfaction over time | Throughout the postoperative examinations (at each follow-up 3 months, 1 year, 3 years, 5 years postoperative)
  The satisfaction of the patient with the spine intervention is evaluated at all postoperative examinations
Return to work status | Throughout the postoperative examinations (at each follow-up 3 months, 1 year, 3 years, 5 years postoperative)

CONTACTS AND LOCATIONS:
Locations (1):
- BG Unfallklinik Frankfurt am Main, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No